CLINICAL TRIAL: NCT00567814
Title: A Double-Blind, Randomized, Placebo-Controlled Study of the Safety and Efficacy of Two Dose Combinations of Metyrapone and Oxazepam in the Treatment of Cocaine Addiction
Brief Title: A Placebo-Controlled Study of a Combination of Metyrapone and Oxazepam in Cocaine Addiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Embera NeuroTherapeutics, Inc. (Industry)
Responsible Party: Marie Lindner, MD/Medical Monitor, Embera NeuroTherapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECA-001
Record Dates: First submitted 2007-12-03; First posted 2007-12-05 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-12

CONDITIONS: Cocaine Dependence; Cocaine Addiction
Keywords: Cocaine; Dependence; Addiction; Cortisol; GABA
MeSH Terms: conditions — Cocaine-Related Disorders; Behavior, Addictive | interventions — Metyrapone; Oxazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Lower dose combination of metyrapone with oxazepam
  Interventions: Drug: Metyrapone; Drug: Oxazepam
- 2 (Active Comparator): Higher dose combination of metyrapone with oxazepam
  Interventions: Drug: Metyrapone; Drug: Oxazepam
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metyrapone — Twice daily
  Other Names: Metopirone
  Arms: 1; 2
Drug: Oxazepam — Twice Daily
  Other Names: Serax
  Arms: 1; 2
Drug: Placebo — Twice daily
  Arms: 3

SUMMARY:
Subjects will be randomly assigned to receive either one of the two potential dose combinations of the study medications or placebo over 6 weeks. The study will include twice weekly visits to the research clinic for laboratory studies, safety assessments and urine drug screens. Subjects will also be questioned regarding drug craving and mood symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 - 50 years of age
* Requests treatment for cocaine addiction
* Meets the DSM-IV criteria for cocaine dependency
* Able to provide written informed consent and comply with the study
* Females of childbearing potential must have a negative pregnancy test and must be using adequate birth control during the study
* Test positive for cocaine on a urinary drug screen
* Healthy and medically stable in the opinion of the Principal Investigator

Exclusion Criteria:

* Liver enzymes greater than two times normal
* Any history of hepatitis
* History of disorders requiring chronic treatment with steroids
* Significantly abnormal ECG
* Any prominent DSM-IV axis I disorders other than cocaine dependence
* Any subject who presents as a danger to self or others in the opinion of the Principal Investigator
* Concomitant use of methamphetamine as determined by self-reporting and verified by measurement of methamphetamine in urinary drug screen
* Alcohol consumption greater than 4 drinks per day (1 Drink = 12 oz beer; 5 oz wine; 1.5 oz shot of liquor)
* Any clinically significant laboratory test abnormalities
* Use of any concomitant medication during the study that would interfere with study medications
* Serum cortisol less than 3 µg/dl at any time before or during study
* Treatment with an investigational product within 30 days prior to study enrollment
* Currently seeking other forms of professional addiction treatment
* Known allergic reaction to oxazepam or metyrapone
* Lactose intolerance

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Reduction or elimination of cocaine craving as evidenced by the Cocaine Craving Questionnaire | 6 weeks

SECONDARY OUTCOMES:
Reduction or elimination of cocaine use as evidenced by self-report and urine toxicology | 6 weeks
Improvement in anxiety and depression symptoms | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anita S Kablinger, MD, Principal Investigator — LSU Health Sciences Center - Shreveport
Locations (1):
- Department of Psychiatry, Psychopharmacology Research Clinic, Shreveport, Louisiana, United States